CLINICAL TRIAL: NCT01659151
Title: A Phase II Clinical Trial of Vemurafenib With Lymphodepletion Plus Adoptive Cell Transfer and High Dose IL-2 in Patients With Metastatic Melanoma
Brief Title: Vemurafenib With Lymphodepletion Plus Adoptive Cell Transfer & High Dose IL-2 Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16992
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Results first posted 2022-02-03 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Melanoma
Keywords: metastatic; melanoma; cell transfer; ACT; T-cell; immunotherapy; antibodies; lymphocytes
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Interleukin-2; aldesleukin; Vemurafenib; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Therapy (Experimental): Combination Chemotherapy and Immunotherapy. The combination of vemurafenib followed by lymphodepletion with chemotherapy, Adoptive Cell Therapy (ACT) with Tumor Infiltrating Lymphocytes (TIL) infusion, and High Dose Interleukin-2 (IL-2).
  Interventions: Drug: High Dose Interleukin-2 (IL-2); Procedure: ACT with TIL Infusion; Drug: Vemurafenib; Drug: Lymphodepletion

INTERVENTIONS:
Drug: High Dose Interleukin-2 (IL-2) — A high dose regimen of IL-2 will be given after participants receive the infusion of the T-cells.
  Other Names: aldesleukin; Proleukin
Procedure: ACT with TIL Infusion — Special immune T-cells will be taken from a sample of the participant's tumor tissue that will be surgically removed. Certain parts of these cells will be multiplied, or grown, in the laboratory. They will then be given back to the participant by an infusion in their veins. These cells are called tumor infiltrating lymphocytes (TIL).
Drug: Vemurafenib — Vemurafenib is used to slow the growth of certain types of cancer cells. This drug will be given for about 3 weeks while T-cells are being grown in the lab and then again after T-cell infusion for up to 2 years.
  Other Names: Zelboraf; B-Raf enzyme inhibitor
Drug: Lymphodepletion — The purpose of lymphodepletion in this study is to temporarily reduce the number of normal lymphocytes circulating in the participant's body before they are given the T-cells that were grown in the lab. This is so that there will be more "space" for the lymphocytes (T-cells) that will be infused in their veins. Fludarabine and cyclophosphamide, 2 types of chemotherapy drugs will be used for what is called lymphodepletion.
  Other Names: fludarabine; Fludara; cyclophosphamide; Neostar; Cytoxan

SUMMARY:
The purpose of this study is to find out more about the effects of an investigational combination of medicines, which includes special immune cells (T-cells).

A T-cell is a type of lymphocyte, or white blood cell. Lymphocytes are a kind of white blood cell that protect the body from viral infections, help other cells fight bacterial and fungal infections, produce antibodies, fight cancers, and coordinate the activities of other cells in the immune system.

DETAILED DESCRIPTION:
In this study, these special immune T-cells will be taken from a sample of the participant's tumor tissue that will be surgically removed. Certain parts of these cells will be multiplied, or grown, in the laboratory. They will then be given back to the patient by an infusion in their veins. These cells are called tumor infiltrating lymphocytes (TIL). The investigators want to study the benefits and side effects of TIL when they are given with the following combination of drugs:

* Vemurafenib - a type of drug used to slow the growth of certain types of cancer cells. This drug will be given for about three weeks while T-cells are being grown in the lab and then again after T-cell infusion for up to two years.
* Fludarabine and cyclophosphamide - two types of chemotherapy drugs. These drugs will be used for what is called lymphodepletion. The purpose of lymphodepletion in this study is to temporarily reduce the number of normal lymphocytes circulating in the patient's body before they are given the T-cells that were grown in the lab. This is so that there will be more "space" for the lymphocytes (T-cells) that will be infused in their veins.
* Interleukin-2 (IL-2) - a drug used to help the body's response to treatment on the immune system. A high dose regimen of IL-2 will be given after they receive the infusion of the T-cells.

The use of TIL is investigational, meaning it has not been approved by the U.S. Food and Drug Administration (FDA). Vemurafenib and IL-2 have been approved by the FDA for the treatment of metastatic melanoma and melanoma that cannot be surgically removed. The chemotherapy drugs fludarabine and cyclophosphamide, used for lymphodepletion, have been approved by the FDA, but not for the treatment of metastatic melanoma.

The combination of vemurafenib followed by lymphodepletion with chemotherapy, TIL infusion, and high dose IL-2 is investigational, and has not been proven to help treat melanoma. This combination is not FDA approved; however, the FDA is allowing its use in this study.

ELIGIBILITY:
Inclusion Criteria:

* Must have unresectable metastatic stage IV melanoma or stage III intransit or regional nodal disease and in the opinion of the PI or treating Coinvestigator is an acceptable candidate for adoptive cell transfer (ACT).
* Residual measurable disease after resection of target lesion(s) for TIL growth
* Tumor must have a B-RAF V600E, D or K mutation by pyrosequencing, Cobas assay, or equivalent (43)
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 - 1. ECOG performance status of 0-1 will be inferred if the patient's level of energy is ≥ 50% of baseline.
* May be treatment-naïve or may have been previously treated for metastatic disease.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of starting Vemurafenib.
* Adequate renal, hepatic and hematologic function, including creatinine of less than or equal to 1.7 gm/dL, total bilirubin less than or equal to 2.0 mg/dL, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dL, aspartic transaminase (AST) and alanine transaminase (ALT) of less than 3X institutional upper limit of normal, hemoglobin of 8 gm/dL or more, white blood count (WBC) of 3000 per mcL and total granulocytes of 1000 per mcL or more, and platelets of 100,000 per mcL or more.
* Must have a positive screening Epstein-Barr Virus (EBV) antibody titre on screening test
* Patients with antibiotic allergies per se are not excluded; although the production of TIL for adoptive transfer includes antibiotics, extensive washing after harvest will minimize systemic exposure to antibiotics.
* At screening, patients with ≤ 3 untreated CNS metastases may be included provided none of the untreated lesions are > 1 cm in greatest dimension, and there is no peri-tumoral edema present on brain imaging (MRI or CT if MRI is contraindicated).
* At screening, patients with ≤ 3 treated central nervous system (CNS) metastases treated with either surgical resection and/or radiation therapy may be included. Patients may be included if the largest lesion is ≤ 1 cm, and there is no evidence of progressive CNS disease on brain imaging at least 28 days after treatment.
* At screening, may be included if the largest lesion is > 1 cm or > 3 in number, and there is no evidence of progressive CNS disease on brain imaging at least 90 days after treatment with surgery and/or radiation therapy.
* At screening, must have no known history of congenital long QT syndrome and must have a corrected mean QTc interval ≤ 450 msec at baseline.
* No evidence of ongoing cardiac dysrhythmia ≥ grade 2, NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0
* All laboratory and imaging studies must be completed and satisfactory within 30 days of signing the consent document, with the exceptions of: negative serum pregnancy test for WOCBP must be negative within 7 days of starting Vemurafenib, human leukocyte antigen (HLA) typing which will not be repeated if performed previously, and pulmonary function tests/cardiac stress tests whose results are valid for 6 months if performed previously.

Exclusion Criteria:

* Patients with active systemic infections requiring intravenous antibiotics, coagulation disorders or other major medical illness of the cardiovascular, respiratory or immune system, which in the opinion of the principal investigator (PI) or treating co-investigator is not acceptable risk for ACT, are excluded.
* Patients testing positive for HIV titre, Hepatitis B surface antigen, Hepatitis B core antibody, Hepatitis C antibody, human T-cell lymphotropic virus type (HTLV) I or II antibody, or both rapid plasma reagin (RPR) and fluorescent treponemal antibodies (FTA) positive
* Patients who are pregnant or nursing
* Patients needing chronic, immunosuppressive systemic steroids are excluded
* Patients with autoimmune diseases that require immunosuppressive medications
* Presence of a significant psychiatric disease, which in the opinion of the principal investigator or his designee, would prevent adequate informed consent or render immunotherapy unsafe or contraindicated
* Patients with > 3 untreated CNS metastases or evidence of peri-tumoral edema
* Patients with ≤ 3 untreated CNS metastases but with at least one lesion >1 cm or peri-tumoral edema
* Patients with congenital long QT syndrome
* Patients with invasive malignancy other than melanoma at the time of enrollment and within 2 years prior to the first Vemurafenib administration are excluded, except for adequately treated (with curative intent) basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix, in situ ductal adenocarcinoma of the breast, in situ prostate cancer, or limited stage bladder cancer or other cancers from which the patient has been disease-free for at least 2 years.
* Unable to swallow pills
* Patients with treated CNS metastases > 1 cm or > 3 in number will be excluded if there is evidence of progressive CNS disease on brain imaging at least 90 days after treatment with surgery and/or radiation therapy.
* Unable to comprehend and give informed consent
* Previous BRAF inhibitor treatment
* Male patients with female partners of childbearing potential who do not agree to use 2 FDA-accepted forms of contraception during sexual intercourse with women of child-bearing potential from the start of Vemurafenib and up to at least 6 months after discontinuing Vemurafenib
* WOCBP who do not agree to use 2 FDA forms of contraception during sexual intercourse from the start of Vemurafenib and up to at least 6 months after discontinuing Vemurafenib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-08-03 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2025-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amod Sarnaik, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Therapy
Started | 17
Completed | 16
Not Completed | 1
Not completed — Inadequate TIL growth | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combination Therapy
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response (OR)
Description: Overall response (OR) is defined as the patient being alive at month 12, and tumor size evaluated at screening and at month 12 using the RECIST 1.1 criteria to be a complete response (CR) or partial response (PR). Evaluations will be made by CT scan approximately 12 months from the date of tumor harvest, and by clinical evaluation during the first 12 months
Time Frame: 12 Months
Population: Evaluable participants
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 16
percentage of participants | 38

2. Primary Outcome: Percentage of Participant Drop Out Rate
Description: The percentage of participants who drop out due to progression between the time of harvest and TIL transfer (i.e., the "drop-out rate").
Time Frame: Up to 12 months
Population: Evaluable participants
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 16
percentage of participants | 6

3. Secondary Outcome: Number of Participants With Progression Free Survival (PFS)
Description: Progression-free survival (PFS), defined as the time from study entry to disease progression, relapse or death due to any cause, whichever is earlier, will be summarized with the Kaplan-Meier curve. Confidence intervals for the median and survival rates at different time points will be constructed if needed and appropriate. This secondary endpoint will be reported descriptively.
Time Frame: 12 months
Population: Evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 16
Participants | 7

ADVERSE EVENTS:
Time Frame: 6 months after end of last treatment, an average of 17 months
Arm/Group | Combination Therapy
All-Cause Mortality (participants affected / at risk) | 4/17
Serious Adverse Events (participants affected / at risk) | 13/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=17)
Intracranial Hemorrhage (Nervous system disorders) | 2 (4)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (10)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (3)
Fever (General disorders) | 1 (1)
Death - NOS (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify - anasarca (General disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Delirium (Psychiatric disorders) | 1 (1)
Immune system disorders - Other, specify - guillian barre syndrome (Immune system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=17)
Nausea (Gastrointestinal disorders) | 16 (45)
Vomiting (Gastrointestinal disorders) | 11 (25)
Diarrhea (Gastrointestinal disorders) | 10 (22)
Constipation (Gastrointestinal disorders) | 6 (11)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 6 (6)
Mucositis oral (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Dry Mouth (Gastrointestinal disorders) | 4 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Bloating (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 16 (25)
Fatigue (General disorders) | 16 (40)
General disorders and administration site conditions - Other, specify (General disorders) | 8 (11)
Pain (General disorders) | 8 (13)
Edema Limbs (General disorders) | 7 (11)
Non-cardiac chest pain (General disorders) | 6 (11)
Localized edema (General disorders) | 5 (5)
Fever (General disorders) | 4 (11)
Flu like symptoms (General disorders) | 3 (3)
Malaise (General disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 16 (108)
Neutrophil count decreased (Investigations) | 16 (47)
Platelet count decreased (Investigations) | 16 (81)
White blood cell decreased (Investigations) | 15 (78)
Alanine aminotransferase increased (Investigations) | 12 (36)
Alkaline phosphatase increased (Investigations) | 12 (36)
Aspartate aminotransferase increased (Investigations) | 10 (19)
Electrocardiogram QT corrected interval prolonged (Investigations) | 7 (15)
Blood bilirubin increased (Investigations) | 5 (18)
Creatinine increased (Investigations) | 5 (7)
Lymphocyte count increased (Investigations) | 2 (2)
Cardiac troponin T increased (Investigations) | 1 (2)
Cholesterol high (Investigations) | 1 (1)
CPK increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (3)
Urine output decreased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (2)
Weight loss (Investigations) | 1 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 16 (47)
Hypophosphatemia (Metabolism and nutrition disorders) | 15 (38)
Hypocalcemia (Metabolism and nutrition disorders) | 13 (30)
Anorexia (Metabolism and nutrition disorders) | 12 (21)
Hyponatremia (Metabolism and nutrition disorders) | 11 (30)
Hypermagnesemia (Metabolism and nutrition disorders) | 7 (12)
Hypokalemia (Metabolism and nutrition disorders) | 6 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (5)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (18)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (38)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 11 (30)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (12)
Photosensitivity (Skin and subcutaneous tissue disorders) | 7 (11)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (13)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (6)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 16 (101)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (15)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (42)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 15 (32)
Dizziness (Nervous system disorders) | 5 (9)
Dysgeusia (Nervous system disorders) | 5 (5)
Presyncope (Nervous system disorders) | 3 (3)
Intracranial hemorrhage (Nervous system disorders) | 2 (4)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (6)
Paresthesia (Nervous system disorders) | 2 (3)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (17)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 13 (21)
Palpitations (Cardiac disorders) | 5 (8)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 5 (5)
Upper respiratory infection (Infections and infestations) | 4 (6)
Urinary tract infection (Infections and infestations) | 3 (3)
Papulopustular rash (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 2 (9)
Eye infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Salivary gland infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Blurred vision (Eye disorders) | 7 (9)
Eye disorders - Other, specify (Eye disorders) | 5 (6)
Photophobia (Eye disorders) | 3 (3)
Conjunctivitis (Eye disorders) | 2 (3)
Dry eye (Eye disorders) | 2 (2)
Floaters (Eye disorders) | 2 (2)
Uveitis (Eye disorders) | 2 (2)
Eye pain (Eye disorders) | 1 (1)
Flashing lights (Eye disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 6 (6)
Hypertension (Vascular disorders) | 6 (7)
Hypotension (Vascular disorders) | 5 (6)
Hot flashes (Vascular disorders) | 4 (4)
Flushing (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (9)
Anxiety (Psychiatric disorders) | 5 (5)
Delirium (Psychiatric disorders) | 2 (3)
Depression (Psychiatric disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 5 (5)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 4 (5)
Seroma (Injury, poisoning and procedural complications) | 4 (4)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (2)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (11)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (15)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 2 (2)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 4 (4)
Hematuria (Renal and urinary disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (2)
Renal calculi (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 4 (5)
Allergic reaction (Immune system disorders) | 1 (2)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1)
Menopause (Social circumstances) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT01659151/Prot_SAP_000.pdf